CLINICAL TRIAL: NCT04299321
Title: LAMA2 Retrospective Review of Medical Charts in Infants & Toddlers With LAMA2-Congenital Muscular Dystrophy
Brief Title: Retrospective Natural History Study of Infants and Toddlers With LAMA2-CMD
Acronym: LAMA2 rNHS
Status: Completed | Type: Observational
Sponsor: Prothelia, Inc. (Industry)
Collaborators: Cure CMD (Other); The Bönnemann Laboratory, NINDS, National Institutes of Health (Unknown); Children's Hospital of Philadelphia (Other); The Beggs Laboratory, Boston Children's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRO-LAMA2-001
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Merosin Deficient Congenital Muscular Dystrophy
Keywords: LAMA2; LAMA2-CMD; CMD; MDC1A; LAMA2-MD; Merosin Deficient
MeSH Terms: conditions — Muscular dystrophy congenital, merosin negative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective chart review study of 75-120 LAMA2-CMD patients will expand the investigators understanding of the natural history of this disease. Current and pending publications cover research performed only in ages 5-16 years; there is currently no documented natural history for patients ages 0-5 years. Data collected in this study has the potential to inform the design of future interventional studies that draw nearer to clinical trial readiness every day.

DETAILED DESCRIPTION:
LAMA2-related congenital muscular dystrophy (LAMA2-CMD) is caused by a deficiency of the α2 subunit of laminin due to mutation of the LAMA2 gene.

Typical LAMA2-CMD cases present with prominent hypotonia and weakness in infancy. Congenital contractures are a common finding in the hands and feet. Weakness and contractures are slowly progressive, and most patients do not achieve independent ambulation. Facial weakness and jaw contractures disrupt normal feeding, resulting in failure to thrive. Most patients require nutrition support at an early age. Cardiac involvement is rare. In addition to neuromuscular aspects of the disorder, patients with LAMA2-CMD have central nervous system findings including prominent T2 and fluid-attenuated inversion recovery (FLAIR) abnormalities in the white matter on brain MRI. Despite the prominent changes on MRI, cognitive function is normal, although patients are at risk of seizures, which are seen in 30% of patients.

A number of potential therapies are currently in development for LAMA2-CMD. A larger prospective natural history was conducted at the National Institutes of Health in LAMA2-CMD patients, ages 5-16 years of age, testing and validating a wide variety of outcome measures suitable for use in clinical trials. However, appropriate clinical outcome measures in younger patients (ages 0-5 years) have yet to be validated.

Some treatments currently in development will almost certainly be more effective the earlier the treatment is administered. Given that there is a distinct lack of data for affected individuals less than 6 years of age, this study will be instrumental in building outcome measures appropriate in younger patients. In order to obtain regulatory authorization to launch clinical trials in affected individuals less than 6 years of age, a documented natural history for this age group must be demonstrated.

The primary objective of this study is to characterize aspects of LAMA2-CMD in ages 0-5 years through medical chart review/data extraction, and participant survey. This study aims to derive clinical trial endpoints useful in conducting interventional trials in the near future.

The secondary objectives of this study include identifying potential prognostic variables of LAMA2-CMD, identifying adverse events associated with LAMA2-CMD that warrant monitoring and potential preventative measures, and to grow the knowledge base of care standards and optimization to improve the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with LAMA2-CMD through:

   1. genetic confirmation of two (2) pathogenic mutations in LAMA2 -OR-
   2. genetic confirmation of one (1) pathogenic mutation in LAMA2, and supporting clinical phenotype based on two or more of the following: physical examination, brain imaging, muscle imaging, muscle biopsy, and creatine kinase (CK) levels (blood test)
2. Patients may be living or deceased
3. Patients may be male or female
4. Patients with available medical records between 2000-2017, documenting diagnosis, observation, and treatment between ages 0-5 years and a minimum set of data covering 12-24 months during this age period.
5. Patients with medical charts available in English
6. Patients (or Parents of minor patients) who are able to consent to participation in English or Spanish, either directly, or through their own trusted interpreter
7. Patients between the ages of 8-17 years who are able to provide assent to participation in English or Spanish, either directly, or through their own trusted interpreter

Exclusion Criteria:

1. Patients not diagnosed with LAMA2-CMD
2. Patients with no available medical records documenting diagnosis, observation, and treatment between ages 0-5 years
3. Patients with medical charts not available in English
4. Patients (or Parents of minor patients) not able to consent to participation in English or Spanish, either directly, or through their own trusted interpreter

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants and toddlers affected by LAMA2-CMD
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To characterize the natural history of LAMA2-CMD | Birth to 5 years of age
  To characterize aspects of LAMA2-CMD in ages 0-5 years through medical chart review/data extraction, and participant survey. This study aims to derive clinical trial endpoints useful in conducting interventional trials in the near future.

SECONDARY OUTCOMES:
To identify potential prognostic variables of LAMA2-CMD | Birth to 5 years of age
  Overall analysis
To identify disease symptoms associated with LAMA2-CMD that warrant monitoring and potential preventative measures | Birth to 5 years of age
  Overall analysis

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bönnemann, MD, Study Director — NINDS/NIH; Reghan Foley, MD, Study Director — NINDS/NIH; Oscar H Mayer, MD, Study Director — Children's Hospital of Philadelphia; Alan Beggs, PhD, Study Director — Boston Children's Hospital; Gustavo Dziewczapolski, PhD, Principal Investigator — Cure CMD; Rachel Alvarez, BS, Study Director — Cure CMD
Locations (1):
- Cure CMD, Inc., Lakewood, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will shared in a peer-reviewed publication. De-identified data will be used to inform future studies.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available indefinitely through publication in approximately 18 months (August 2021)
Access Criteria: Journal will have free access through PubMed

REFERENCES:
- [Background] Foley AR, Quijano-Roy S, Collins J, Straub V, McCallum M, Deconinck N, Mercuri E, Pane M, D'Amico A, Bertini E, North K, Ryan MM, Richard P, Allamand V, Hicks D, Lamande S, Hu Y, Gualandi F, Auh S, Muntoni F, Bonnemann CG. Natural history of pulmonary function in collagen VI-related myopathies. Brain. 2013 Dec;136(Pt 12):3625-33. doi: 10.1093/brain/awt284. Epub 2013 Nov 22. PMID 24271325
- [Background] Nadeau A, Kinali M, Main M, Jimenez-Mallebrera C, Aloysius A, Clement E, North B, Manzur AY, Robb SA, Mercuri E, Muntoni F. Natural history of Ullrich congenital muscular dystrophy. Neurology. 2009 Jul 7;73(1):25-31. doi: 10.1212/WNL.0b013e3181aae851. PMID 19564581
- [Background] Ditaranto R, Boriani G, Biffi M, Lorenzini M, Graziosi M, Ziacchi M, Pasquale F, Vitale G, Berardini A, Rinaldi R, Lattanzi G, Potena L, Martin Suarez S, Bacchi Reggiani ML, Rapezzi C, Biagini E. Differences in cardiac phenotype and natural history of laminopathies with and without neuromuscular onset. Orphanet J Rare Dis. 2019 Nov 19;14(1):263. doi: 10.1186/s13023-019-1245-8. PMID 31744510
- [Background] Durbeej M. Laminin-alpha2 Chain-Deficient Congenital Muscular Dystrophy: Pathophysiology and Development of Treatment. Curr Top Membr. 2015;76:31-60. doi: 10.1016/bs.ctm.2015.05.002. PMID 26610911
- [Background] Jain MS, Meilleur K, Kim E, Norato G, Waite M, Nelson L, McGuire M, Duong T, Keller K, Lott DJ, Glanzman A, Rose K, Main M, Fiorini C, Chrismer I, Linton M, Punjabi M, Elliott J, Tounkara F, Vasavada R, Logaraj R, Winkert J, Donkervoort S, Leach M, Dastgir J, Hynan L, Nichols C, Hartnett E, Averion GM, Collins JC, Kim ES, Kokkinis A, Schindler A, Zukosky K, Fee R, Hinton V, Mohassel P, Bharucha-Goebel D, Vuillerot C, McGraw P, Barton M, Fontana J, Rutkowski A, Foley AR, Bonnemann CG. Longitudinal changes in clinical outcome measures in COL6-related dystrophies and LAMA2-related dystrophies. Neurology. 2019 Nov 19;93(21):e1932-e1943. doi: 10.1212/WNL.0000000000008517. Epub 2019 Oct 25. PMID 31653707
- [Background] Bendixen RM, Butrum J, Jain MS, Parks R, Hodsdon B, Nichols C, Hsia M, Nelson L, Keller KC, McGuire M, Elliott JS, Linton MM, Arveson IC, Tounkara F, Vasavada R, Harnett E, Punjabi M, Donkervoort S, Dastgir J, Leach ME, Rutkowski A, Waite M, Collins J, Bonnemann CG, Meilleur KG. Upper extremity outcome measures for collagen VI-related myopathy and LAMA2-related muscular dystrophy. Neuromuscul Disord. 2017 Mar;27(3):278-285. doi: 10.1016/j.nmd.2016.11.017. Epub 2016 Dec 5. PMID 28087121
- [Background] Fauroux B, Amaddeo A, Quijano-Roy S, Barnerias C, Desguerre I, Khirani S. Respiratory insight to congenital muscular dystrophies and congenital myopathies and its relation to clinical trial. Neuromuscul Disord. 2018 Sep;28(9):731-740. doi: 10.1016/j.nmd.2018.06.013. Epub 2018 Jul 1. PMID 30097248
- [Background] Wicklund MP. Rare disease clinical trials: Power in numbers. Neurol Genet. 2016 Aug 4;2(4):e92. doi: 10.1212/NXG.0000000000000092. eCollection 2016 Aug. PMID 27540592
- [Result] Butterfield RJ. Congenital Muscular Dystrophy and Congenital Myopathy. Continuum (Minneap Minn). 2019 Dec;25(6):1640-1661. doi: 10.1212/CON.0000000000000792. PMID 31794464
- [Result] Meilleur KG, Jain MS, Hynan LS, Shieh CY, Kim E, Waite M, McGuire M, Fiorini C, Glanzman AM, Main M, Rose K, Duong T, Bendixen R, Linton MM, Arveson IC, Nichols C, Yang K, Fischbeck KH, Wagner KR, North K, Mankodi A, Grunseich C, Hartnett EJ, Smith M, Donkervoort S, Schindler A, Kokkinis A, Leach M, Foley AR, Collins J, Muntoni F, Rutkowski A, Bonnemann CG. Results of a two-year pilot study of clinical outcome measures in collagen VI- and laminin alpha2-related congenital muscular dystrophies. Neuromuscul Disord. 2015 Jan;25(1):43-54. doi: 10.1016/j.nmd.2014.09.010. Epub 2014 Sep 28. PMID 25307854